CLINICAL TRIAL: NCT06776224
Title: Evaluation of Neuroaxonal Loss Outside of Any Inflammation in Multiple Sclerosis by a Multimodal Study of the Visual Pathways Model
Brief Title: Visual (Path)Ways in Multiple Sclerosis - Part II
Acronym: VWIMS - II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024_0018; 2024-A01517-40 (Other: IDRCB)
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis, Optic Neuritis, Demyelinating Disease
Keywords: Multiple sclerosis, cognition, OCT, MRI, visual impairment
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis; Demyelinating Diseases; Ornithine Carbamoyltransferase Deficiency Disease; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Not applicable. No treatment will be compared. (Other): During the same visit, we will perform OCT-angiography (10 minutes) and evaluate visual cognition with an eye-tracker (20 minutes)
  Interventions: Other: Measurement of retinal vascular density and visual cognition

INTERVENTIONS:
Other: Measurement of retinal vascular density and visual cognition — During the same visit, we will perform OCT-angiography (10 minutes) and evaluate visual cognition with an eye-tracker (20 minutes)

SUMMARY:
Multiple sclerosis (MS) is an inflammatory demyelinating and degenerative disease of the central nervous system. The mechanisms of neuro-axonal loss remain incompletely elucidated. An acute demyelinating lesion will produce both immediate and delayed axonal loss. Immediate axonal loss is linked to the occurrence of axonal transection. Delayed axonal loss is the cause of axonal degeneration in progressive MS. Visual impairment is common in the disease (vision, oculomotricity, cognition). Through a longitudinal multimodal analysis of visual pathways, we would like to investigate physiopathological mechanisms leading to neurodegenerative process and visual impairment.

ELIGIBILITY:
Patients with relapsing-remitting multiple sclerosis receiving high-efficacy or non-high-efficacy treatment and follow-up at the CRCSEP of the Lille University Hospital through past participation in the VWIMS study.

Inclusion criteria:

* Male and/or female participants in the VWIMS research project
* At least 18 years of age at the time of inclusion in VWIMS - II
* Patient having given written consent to participate in the study
* Socially insured patient
* Patient willing to comply with all study procedures and duration

Exclusion Criteria:

* Age < 18 years
* Other neurological pathologies that may interfere with MRI and/or OCT data (diabetes, retinopathy [any cause], glaucoma, retinal detachment, ametropia > 6 diopters)
* Contraindications to MRI (claustrophobia, incompatible metal foreign bodies such as certain pacemakers and mechanical valves, cochlear implants, intra-orbital metal splinters, pregnancy, certain brands of IUD because of the 3 Tesla magnetic field).
* Contraindication to injection: severe renal failure with creatine clearance <30, allergy to contrast media, pregnancy, breast-feeding.
* Pregnant women
* Nursing women
* Persons incapable of giving consent on their own, with or without legal protection (guardianship/curatorship)
* Person under legal protection
* Persons deprived of their liberty
* Administrative reasons: inability to receive informed information, inability to participate in the entire study, lack of social security coverage, refusal to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-04-24 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Quantifying progressive retinal axonal loss in the absence of inflammation | First time point already done (VWIMS study) Second time point during VWIMS -II study. Interval between time points will be around 7-8 years
  To quantify progressive retinal neuroaxonal loss in a context of no active inflammation : Difference in retinal atrophy (GCIPL volume in [VWIMS I] - GCIPL volume in VWIMS II)

CONTACTS AND LOCATIONS:
Locations (1):
- Direction de la Recherche et de l'innovation (DRI) 6 rue Professeur Laguesse, Lille, France